CLINICAL TRIAL: NCT05794503
Title: Postoperative Urinary Retention After Reversal of Neuromuscular Block by Neostigmine Versus Sugammadex in Patients Undergoing Laparoscopic Cholecystectomy: A Randomized Controlled Trial
Brief Title: Postoperative Urinary Retention After Reversal of Neuromuscular Block by Neostigmine Versus Sugammadex
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Tiffany B Moon, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU-2022-1201
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-09

CONDITIONS: Urinary Retention Postoperative; Laparoscopic Cholecystectomy; Neuromuscular Blockade; Sugammadex; Neostigmine; Neuromuscular Blocking Agents; Physiological Effects of Drugs
MeSH Terms: interventions — Neostigmine; Sugammadex

STUDY DESIGN:
Intervention Model Description: Single site, randomized, controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Neostigmine (Active Comparator): One type of Neuromuscular Blockade Reversal Drug
  Interventions: Drug: Neostigmine
- Sugammadex (Active Comparator): One type of Neuromuscular Blockade Reversal Drug
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Neostigmine — Maintenance neuromuscular blockade with boluses of rocuronium. For reversal, neostigmine.
  Arms: Neostigmine
Drug: Sugammadex — Maintenance neuromuscular blockade with boluses of rocuronium. For reversal, sugammadex
  Arms: Sugammadex

SUMMARY:
This study is intended to be a single-site, prospective, randomized, controlled study that intends to enroll a total of 230 patients undergoing laparoscopic cholecystectomy at Parkland Hospital. Patients will be randomized to receive either neostigmine or sugammadex for reversal of rocuronium-induced neuromuscular blockade. A standardized anesthetic protocol that is usual and customary for the type of operation the patient is having will be provided to the anesthesia teams of enrolled subjects. The remainder of the anesthetic care of the subject will not deviate from the standard of care. To account for protocol deviations and patient dropout, up to 250 randomization envelopes will be made and enrollment will continue until there are 230 completed enrollments.

DETAILED DESCRIPTION:
Objective:

To determine the incidence of postoperative urinary retention after reversal of rocuronium-induced neuromuscular blockade by neostigmine versus sugammadex in patients undergoing laparoscopic cholecystectomy.

Hypothesis:

Subjects who are reversed with sugammadex will have less postoperative urinary retention compared to subjects who are reversed with neostigmine.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old
* Undergoing laparoscopic cholecystectomy
* Anticipated surgical duration <2 hours
* ASA physical status classification 1-3
* Willing and able to consent in English or Spanish
* No personal history of neuromuscular disease

Exclusion Criteria:

* Preoperative urinary catheter
* History of problems with urination
* Current use of anticholinergic medications (e.g., antihistamines, phenothiazines, antidepressants, antipsychotics)
* Current UTI or urogenital problem (incontinence, known bladder retention, prostate hypertrophy)
* Planned intraoperative insertion of a urinary catheter
* ESRD (GRF <30 mL/min)
* ESLD (AST or ALT > 3x reference range)
* Planned postoperative intubation/ventilation or admission to ICU
* Allergy to sugammadex, neostigmine, glycopyrrolate, or rocuronium
* Pregnant or nursing women
* "Stat" (emergent) cases
* Known or suspected neurological condition (e.g., Alzheimer's, h/o of stroke, multiple sclerosis, Parkinson's)
* Patients on toremifene (a selective estrogen receptor modulator)
* Women on oral contraceptives who do not wish to use a non-hormonal method of contraception for 7 days following surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Moon, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neostigmine | Sugammadex
Started | 117 | 118
Completed | 112 | 118
Not Completed | 5 | 0
Not completed — Operation Cancelled | 2 | 0
Not completed — Received Neostigmine + Sugammadex | 2 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neostigmine | Sugammadex | Total
Number analyzed (Participants) | 112 | 118 | 230
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 106 | 106 | 212
  >=65 years | 6 | 12 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 89 | 176
  Male | 25 | 29 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 103 | 99 | 202
  Not Hispanic or Latino | 9 | 19 | 28
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 112 | 118 | 230

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postoperative Urinary Retention (POUR) of Sugammadex and Neostigmine Groups
Description: Measure pre- and post-void bladder volumes, void volume, and the time to void after operation.
  The count of participants with Postoperative Urinary Retention (POUR) of Sugammadex and Neostigmine Groups is being reported.
  POUR will be defined as:
  1. Inability to spontaneously urinate and a bladder volume ≥ 300 mL
  2. Postvoid residual > 150 mL
  3. Need for insertion of Foley catheter or straight catheter
Time Frame: In the post-operative anesthesia care unit, bladder volumes and time to void were measured, assessed up to 24 hours or patient discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Neostigmine | Sugammadex
Number analyzed (Participants) | 112 | 118
Participants | 20 | 6

ADVERSE EVENTS:
Time Frame: Up to post operative day 30
Arm/Group | Neostigmine | Sugammadex
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/118
Serious Adverse Events (participants affected / at risk) | 0/112 | 0/118
Other Adverse Events (participants affected / at risk) | 0/112 | 0/118

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-05): https://cdn.clinicaltrials.gov/large-docs/03/NCT05794503/Prot_SAP_001.pdf